CLINICAL TRIAL: NCT05178797
Title: Effects of Kinesiology Taping Technique in Post-mastectomy Breast Cancer Related Lymphedema on Swelling, Upper Limb Function, and Strength
Brief Title: Kinesiology Taping Technique in Post-mastectomy Breast Cancer Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSaleem
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-01

CONDITIONS: Post Mastectomy Lymphedema
Keywords: physiotherapy; breast cancer; breast carcinoma
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of groups (A and B) in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: Statistician will also be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K-tapping and exercise (Group A) (Experimental): Group A will be given kinesiology taping technique and exercise therapy
  Interventions: Other: Kinesiology taping technique with exercise therapy
- Compression decongestive therapy (Group B ) (Active Comparator): Group B will be given compression decongestive therapy (manual lymphatic drainage, short stretch bandage and exercise therapy)
  Interventions: Other: Compression decongestive therapy

INTERVENTIONS:
Other: Kinesiology taping technique with exercise therapy — Kinesiology tape is a latex-free fiber that stretches longitudinally & elastic with an acrylic adhesive. It is used to stimulate dermal mechanoreceptors, encourages sensory and mechanical stimuli resulting in reduction of clogging lymphatic flow which limits the circumference of the affected limb in the region where it is applied due to its flexibility and acts over the lymphatic system. However, exercise therapy is systematic movement program to strengthen muscles.
  Arms: K-tapping and exercise (Group A)
Other: Compression decongestive therapy — It consists of two phases: First is the intensive phase (volume reduction phase), in this phase short stretch bandage, manual lymphatic drainage, skincare and exercises will be given for a period of 4 weeks.
  In the second phase (maintenance phase), compression garments and exercises will be given to the patient for maintaining the limb volume or to reduce the risk of lymphedma.
  Arms: Compression decongestive therapy (Group B )

SUMMARY:
Generally, Breast cancer related to lymphedema is commonly found in the female population after mastectomy. It has many complications which affects the normal functions of an individual and quality of life. This randomized control trial will be conducted on patients who are admitted as patients after mastectomy to determine the effects of kinesiology taping technique in post mastectomy breast cancer related lymphedema on swelling, upper limb function and strength.

DETAILED DESCRIPTION:
Generally, Breast cancer related to lymphedema is commonly found in the female population after mastectomy. It has many complications which affects the normal functions of an individual and quality of life. Traditional therapies like compression decongestive therapies and kinesiology taping techniques are used for the management of post mastectomy breast cancer related lymphedema.This randomized control trial will be conducted on patients who are admitted as patients after mastectomy to determine the effects of kinesiology taping technique in post mastectomy breast cancer related lymphedema on swelling, upper limb function and strength. Total 50 patients with post mastectomy who fulfill the inclusion criteria will be selected after taking consent. The subjects will be allocated into two groups through simple random sampling. Subjects ingroup A will be given kinesiology taping technique and exercise therapy whereas; patients in group B will be given compression decongestive therapy (manual lymphatic drainage, short stretch bandage and exercise therapy). All subjects will be assessed using assessment form, upper limb functional index, dynamometer, pinch meter and tape measure. Assessment will be conducted at base line, after 2 & 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 65
* Patient undergoing Unilateral Modified Radical Mastectomy
* Within 1 week post Mastectomy
* Subjects without swelling or with mild swelling

Exclusion Criteria:

* active cancer or disease that might lead to swelling
* subjects taking anticoagulant therapy
* diagnose skin disease and skin allergies
* vascular insufficiency
* sensory impairments
* open wound and scars which have not healed
* Functional limitations of upper limb before mastectomy e.g. adhesive capsulitis.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study condition can be present in female gender only.
Enrollment: 50 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Change form baseline in upper limb function on the upper limb functional index at sixth session | Baseline and 2 weeks
  tI is a questionnaire to quantify the disability in people with upper extremity conditions.The patient gives a score to each of 20 listed activities based on the difficulty in completing the activities. It consists of 20 activities items in which a score range from 0 to 80. Where, 80 score shows a high level of function and 0 shows disability, each activity score is 0 to 4.This measurement is used for upper limb function and self-reported by patient.
Change form baseline in upper limb function on the upper limb functional index at twelfth session | Baseline and 4 weeks
  It is a questionnaire to quantify the disability in people with upper extremity conditions.The patient gives a score to each of 20 listed activities based on the difficulty in completing the activities. It consists of 20 activities items in which a score range from 0 to 80. Where, 80 score shows a high level of function and 0 shows disability, each activity score is 0 to 4.This measurement is used for upper limb function and self-reported by patient.
Change from baseline in upper limb volume on tape measure at sixth session | Baseline and 2 week
  It is a tool used for the arm circumference measurements and to evaluate the degree of lymphedma. The Patient sits on a chair and his arm is flexed to 900. First measure is taken at the wrist and after 10cm proximal to wrist and so on
Change from baseline in upper limb volume on tape measure at sixth session | Baseline and 4 weeks
  It is a tool used for the arm circumference measurements and to evaluate the degree of lymphedma. The Patient sits on a chair and his arm is flexed to 900. First measure is taken at the wrist and after 10cm proximal to wrist and so on
Change from baseline in upper limb strength on dynamometer and pinch meter at sixth session | Baseline and 2 weeks
  It is a measurement tool used in physiotherapy to assess the highest isometric strength of hand grasp and fingers. It consists of a hydraulic system with a changeable handle size. It measures the strength in pounds/square inch (psi
Change from baseline in upper limb strength on dynamometer and pinch meter at twelfth session | Baseline and 4 weeks
  It is a measurement tool used in physiotherapy to assess the highest isometric strength of hand grasp and fingers. It consists of a hydraulic system with a changeable handle size. It measures the strength in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Saleem Agwan, MSAPT, Principal Investigator — Dow University of Health Sciences
Locations (2):
- Pakistan (2):
  - Dr. Ruth K. M. Pfau, Civil Hospital, Karachi, Sindh
  - Sindh Institute Physical Medicine and Redhabilitation, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No